CLINICAL TRIAL: NCT03141970
Title: Randomized, Multicentric, Open Label, Parallel Group Trial to Compare the Efficacy of 6-months Versus 3-months Therapy With Prednisolone for the First Episode of Idiopathic Nephrotic Syndrome in Children Younger Than 4 Years
Brief Title: Prednisolone Trial in Children Younger Than 4 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: NephCure Accelerating Cures Institute (Unknown); University of Michigan (Other); Department of Biotechnology, Government of India (funding agency) (Unknown)
Responsible Party: Principal Investigator, Arvind Bagga, Professor, Department of Pediatrics, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: v1.0; CTRI/2015/06/005939 (Registry Identifier: Clinical Trials Registry-India)
Record Dates: First submitted 2017-03-17; First posted 2017-05-05 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Nephrotic Syndrome
Keywords: Proteinuria Hypoproteinemia Edema Hypoalbuminemia Prednisone
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Prednisolone; Prednisone

STUDY DESIGN:
Intervention Model Description: Multicentric, Parallel group, Open label randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intervention: Prednisolone (Experimental): Drug: 12- Weeks of Prednisolone Therapy Subjects will add an additional 12 weeks of Prednisolone to follow pre-randomization standard of care prednisolone. Post randomization Prednisolone therapy of 30 mg/m2 on alternate days for 4 weeks, 20 mg/m2 on alternate days for 4 weeks, and 10 mg/m2 on alternate days for 4 weeks
  Interventions: Drug: Prednisolone
- No intervention (No Intervention): Subjects will NOT receive 12-weeks of additional Prednisolone therapy following randomization

INTERVENTIONS:
Drug: Prednisolone — Prednisolone for 12 weeks as follows 30 mg/m2 on alternate days for 4 weeks 20 mg/m2 on alternate days for 4 weeks 10 mg/m2 on alternate days for 4 weeks
  Other Names: Prednisone
  Arms: Intervention: Prednisolone

SUMMARY:
This study is a multicentric, randomized, parallel group, open label controlled trial of children age 1 year up to 4 years with new onset, idiopathic nephrotic syndrome. It is designed to test the initial duration of steroid therapy of either 3 month or 6 month total duration. Participants will be randomized to either extend their pre-trial 3 months (12 weeks) of standard of care corticosteroid therapy to add an additional 12 weeks of therapy or to stop therapy. Pre-trial standard of care corticosteroids will include 60 mg/m2/day for 6 weeks followed by 40 mg/m2/day every other day for 6 weeks of prednisolone or equivalent. The trial intervention will therefore be an additional 12 vs 0 weeks of corticosteroids in these children with idiopathic nephrotic syndrome.

DETAILED DESCRIPTION:
Trial Registration Note:This trial was initially registered in the Indian Registry (list the number) on (date) prior to enrolling participants. The present listing shows this status of currently enrolling. New sites in the United States are expected to open within the coming year. At that time the answers to some questions, such as "Studies FDA regulated drug" will change because the basis for FDA regulation will reside on the presence of US sites and the use of US manufactured drug, whereas at this time the drug is not of US manufacture, and the trial is not currently conducted in the United States. This registration is being posted at this time to prepare to meet United States FDAAAA registration requirements.

Nephrotic syndrome is a common renal disorder in children characterized by proteinuria, hypoalbuminemia and edema. The long-term prognosis for steroid-sensitive nephrotic syndrome is excellent for resolution of disease and maintenance of renal function. About 80% patients with steroid-sensitive nephrotic syndrome will relapse one or more times, requiring repeated treatment with corticosteroids. Of these, 50-60% show frequent relapses or steroid dependence and require therapy with long-term corticosteroids and other medications. Patients with multiple relapses are at risk for life-threatening infections, malnutrition and thrombotic episodes. They are also likely to show serious side effects of long-term steroid therapy and those related to use of other medications, including toxicity to bone marrow, gonads, central nervous system and kidneys. Repeated relapses also result in multiple hospitalizations and school absence. Strategies effective in reducing relapse rates and proportion of patients with frequent relapses or steroid dependence shall therefore be extremely valuable in improving the long-term management of nephrotic syndrome.

Based on information from multiple studies that prolonged duration of initial therapy beyond 8-weeks reduced the risk of an early relapse and lowered frequency of subsequent relapses, it is agreed upon that the initial therapy with prednisolone should continue for 12 weeks (3 months), administered daily for a duration of 6 weeks, and then on alternate days for another 6 weeks. However, the optimal dose and duration of corticosteroid therapy remains to be determined. Data from various prospective studies, systematically reviewed in the Cochrane Registry, suggests the beneficial effects of prolongation of treatment beyond 3 months, with benefit seen up to 6-months. However, the advantages of extending therapy from 3- to 6-months are not unambiguous; there are also concerns of the corticosteroid toxicity with the latter regimens. Recent placebo controlled trials reported in 2013, including from this center, suggest that extending initial prednisolone treatment from 3 months to 6 months, with or without an increase in cumulative dose, does not influence the course of disease in children with nephrotic syndrome. However, in the study conducted in India, we found that prolonged therapy was useful in postponing the first relapse, and was associated with an insignificantly decreased risk of frequent relapses, in the subgroup of children younger than 4 years. Since the subgroups were not defined a priori, a prospective study is required to clarify the efficacy of this intervention in young patients.

Further, the lack of clarity regarding disease pathogenesis makes the administration of corticosteroid therapies largely empirical. While clear insight into the pathogenic pathways targeted by prednisolone is lacking, there is some evidence that disease remission is associated with down regulation of T cell activation, altered B-T cell crosstalk, upregulation of T helper type 1(Th1) and/or T regulatory compartments.

This present study proposes to examine the benefits of prolongation of initial therapy of idiopathic nephrotic syndrome from the current standard of 3 to 6 months among children younger than 4-yr-old an onset of disease. Prolongation of treatment at the first episode would have considerable promise, if found effective in reducing future relapses and without concomitant risks of corticosteroid toxicity. The proposal also aims to examine the proportions of T and B lymphocyte subsets in 20 patients with the initial episode of nephrotic syndrome. The evaluation shall be conducted at onset of disease, following prednisolone induced disease remission, and at one year from randomization or at first relapse of the disease to determine differences in the immune profiles at different stages of the disease. Apart from improving our knowledge of pathogenesis of nephrotic syndrome, this approach shall enhance our understanding of the immunological alterations influenced by therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic, steroid-sensitive, first episode of nephrotic syndrome
2. Age 12 months up to 48 months
3. Written informed consent

Exclusion Criteria

1. Nephrotic syndrome known to be secondary to a systemic disorder, e.g., Immunoglobulin A (IgA) nephropathy, systemic lupus erythematosus, Henoch Schonlein purpura, vasculitis, , hepatitis B or Alport syndrome.
2. Persistent estimated glomerular filtration rate (GFR) <75 ml/min/1.73 m2,
3. Therapy with prednisolone for prior episodes of nephrotic syndrome,
4. Therapy with corticosteroids in the past 3 months, in a dose more than 1 mg/kg for >14 days for any other reason,
5. Corticosteroid therapy for initial episode of nephrotic syndrome prior to randomization varying from pre-specified protocol on more than 14 days,
6. Patients who show relapse during the first 3 months of pre-randomization corticosteroid therapy for nephrotic syndrome,
7. Unclear treatment history,
8. Gross hematuria,
9. Patients with initial steroid resistance,
10. Participation in any other drug study during the course of this study.
11. Participation in more than one study without approval from the researchers involved in each study,

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Relapse of nephrotic syndrome during 12 months after randomization | 12 month period following randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome

SECONDARY OUTCOMES:
Number of relapses during 12 months follow up | 12 month period following randomization
  Number of nephrotic syndrome relapses per patient year during the 12-month period following randomization
Time to first relapse (days) | 12 month period following randomization
  Number of days from randomization to occurrence of first relapse
Occurrence of frequent relapses of nephrotic syndrome during 12 months from randomization | 12 month period following randomization
  Proportion of patients with frequent relapses during the 12 months post randomization
Cumulative prednisolone [or corticosteroid equivalent] received during 12 month period from randomization | 12 month period following randomization
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 12 months from randomization
The use of steroid-sparing medications | 12 month period following randomization
  The proportion of patients in each study arm treated with steroid-sparing strategies or medications, e.g., levamisole, cyclophosphamide, mycophenolate mofetil and calcineurin inhibitors
Adverse events during 12-month period after randomization | 12 month period following randomization
  Number and types of adverse events experienced, related or unrelated to corticosteroid use
Change in anthropometry and growth velocity during 12-month period after randomization | 12 month period following randomization
  Changes in standard deviation scores (SDS) for weight, height and body mass index during 12-month period following randomization

OTHER OUTCOMES:
In a subgroup of 20 patients, the proportions of the following cell subsets, at baseline and at 6 and 12 months after randomization and at first relapse | 12 month period following randomization
  Proportions of B (naive, memory, regulatory) and T (cytotoxic, helper 1, helper 2, helper 17, regulatory) cell subsets, as determined by flow cytometric staining for specific surface and intracellular markers
Relapse of nephrotic syndrome during 24 months after randomization | 24 month period following randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome
Number of relapses during 24 months follow up | 24 month period following randomization
  Number of nephrotic syndrome relapses per patient year during the 24-month period
Time to first relapse (days) | 24 month period following randomization
  Number of days from randomization to occurrence of first relapse
Occurrence of frequent relapses of nephrotic syndrome during 24 months from randomization | 24 month period following randomization
  Proportion of patients with frequent relapses during the 24 months post randomization
Cumulative prednisolone [or corticosteroid equivalent] received during 24 month period | 24 month period following randomization
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 24 months from randomization
Relapse of nephrotic syndrome during 12 months after randomization in boys compared to girls | 12 month period following randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome in boys compared to girls
Relapse of nephrotic syndrome during 12 months after randomization in patients <2-yr-old at randomization compared to older patients | 12 month period following randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome in patients <2-yr-old at randomization compared to older patients
Relapse of nephrotic syndrome during 12 months after randomization in Indian patients compared to those in the USA | 12 month period following randomization
  Proportion of patients with one or more relapse(s) of nephrotic syndrome in Indian patients compared to those in the USA
Number of relapses during 12 months follow up in boys compared to girls | 12 month period following randomization
  Number of nephrotic syndrome relapses per patient year during the 12-month period in boys compared to girls
Number of relapses during 12 months follow up in patients <2-yr-old at randomization compared to older patients | 12 month period following randomization
  Number of nephrotic syndrome relapses per patient year during the 12-month period in patients <2-yr-old at randomization compared to older patients
Number of relapses during 12 months follow up in Indian patients compared to those in the USA | 12 month period following randomization
  Number of nephrotic syndrome relapses per patient year during the 12-month period in Indian patients compared to those in the USA
Time to first relapse (days) in boys compared to girls | 12 month period following randomization
  Number of days from randomization to occurrence of first relapse in boys compared to girls
Time to first relapse (days) in patients <2-yr-old at randomization compared to older patients | 12 month period following randomization
  Number of days from randomization to occurrence of first relapse in patients <2-yr-old at randomization compared to older patients
Time to first relapse (days) in Indian patients compared to those in the USA | 12 month period following randomization
  Number of days from randomization to occurrence of first relapse in Indian patients compared to those in the USA
Occurrence of frequent relapses of nephrotic syndrome during 12 months from randomization in boys compared to girls | 12 month period following randomization
  Proportion of patients with frequent relapses during the 12 months post randomization in boys compared to girls
Occurrence of frequent relapses of nephrotic syndrome during 12 months from randomization in patients <2-yr-old at randomization compared to older patients | 12 month period following randomization
  Proportion of patients with frequent relapses during the 12 months post randomization in patients <2-yr-old at randomization compared to older patients
Occurrence of frequent relapses of nephrotic syndrome during 12 months from randomization in Indian patients compared to those in the USA | 12 month period following randomization
  Proportion of patients with frequent relapses during the 12 months post randomization in Indian patients compared to those in the USA
Cumulative prednisolone [or corticosteroid equivalent] received during 12 month period in boys compared to girls | 12 month period following randomization
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 12 months from randomization in boys compared to girls
Cumulative prednisolone [or corticosteroid equivalent] received during 12 month period in patients <2-yr-old at randomization compared to older patients | 12 month period following randomization
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 12 months from randomization in patients <2-yr-old at randomization compared to older patients
Cumulative prednisolone [or corticosteroid equivalent] received during 12 month period in Indian patients compared to those in the USA | 12 month period following randomization
  Total amount of prednisolone [or corticosteroid equivalent] received, as mg/kg/day or mg/m2/day as intervention and for treatment of relapses, during 12 months from randomization in Indian patients compared to those in the USA

CONTACTS AND LOCATIONS:
Overall Officials: Arvind Bagga, MD, Principal Investigator — All India Institute of Medical Sciences, New Delhi, India; Debbie Gipson, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (4):
  - Cedars-Sinai Medical Center, Pediatric IBD & Pediatric Nephrology, Los Angeles, California
  - Stanford University Medical Center, Department of Pediatrics, Division of Nephrology, Stanford, California
  - University of Michigan Department of Pedatric Nephrology, Ann Arbor, Michigan
  - Levine's Children/Carolinas HealthCare System, Charlotte, North Carolina
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Following anonymisation to protect patient identity, data from patients in USA will be pooled and analyzed with that from Indian patients. Data will be available once all subjects have completed the study and data has been analyzed. No interim data analysis will be conducted
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Hahn D, Samuel SM, Willis NS, Craig JC, Hodson EM. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Aug 22;8(8):CD001533. doi: 10.1002/14651858.CD001533.pub7. PMID 39171624
- Available data/document: Study Protocol: CTRI/2015/06/005939 — http://ctri.nic.in/Clinicaltrials/login.php — Contains details of registration of clinical trial prior to recruiting patients in India, at website of Clinical Trials Registry of India